CLINICAL TRIAL: NCT01448941
Title: Arthrodesis Versus Extra-articular Bridge Plating of the First Tarsometatarsal Joint After Acute Lisfranc Injury
Brief Title: Arthrodesis Versus Extra-articular Plate Fixation in Lisfranc Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Are Haukåen Stødle, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206025 (REK-ID)
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2018-04

CONDITIONS: Lisfranc Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary arthrodesis TMT 1 (Active Comparator): Arthrodesis TMT 1 when instability is present. Primary arthrodesis TMT 2 and 3 when instability present
  Interventions: Procedure: Primary arthrodesis; Procedure: Primary arthrodesis TMT 2 and 3
- Temporary extraarticular plate fixation (Experimental): Temporary extraarticular plate fixation of TMT 1 when instability is present. Primary arthrodesis TMT 2 and 3 when instability present
  Interventions: Procedure: Temporary extraarticular plate fixation; Procedure: Primary arthrodesis TMT 2 and 3

INTERVENTIONS:
Procedure: Temporary extraarticular plate fixation — Arm 1: Primary arthrodesis TMT 1 Arm 2: Temporary extraarticular plate fixation TMT 1
  Arms: Temporary extraarticular plate fixation
Procedure: Primary arthrodesis — Primary arthrodesis
  Arms: Primary arthrodesis TMT 1
Procedure: Primary arthrodesis TMT 2 and 3 — Primary arthrodesis TMT 2 and 3 when instability is present

SUMMARY:
The purpose of this study is to compare arthrodesis of the first TMT-joint to extraarticular bridge plate fixation of the same joint in acute Lisfranc injuries.

DETAILED DESCRIPTION:
We want to compare arthrodesis of TMT 1 to temporary bridge plating of TMT 1 in acute Lisfranc injuries where at least tarsometatarsal joints 1-3 are involved.

We preform arthrodesis of TMT 2 and 3 in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Lisfranc injuries with instability off TMT1, and fracture/instability of TMT 2 and 3. No major fracture in relation to TMT1.
* Age 18-65

Exclusion Criteria:

* Feet with other major foot/ankle injuries
* Previous foot infection or foot pathology on affected side
* Previous surgery to the TMT joints
* Sequelae after previous foot injuries
* Diabetes mellitus, neuropathy and peripheral vascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
AOFAS Midfoot scale | 2 years postoperative
  AOFAS Midfoot scale

SECONDARY OUTCOMES:
SF-36 | 2 years postoperative
  SF-36

OTHER OUTCOMES:
ROM TMT 1 after temporary plate fixation | 1 year post operative
  ROM will be measured by Radiosterometric analysis (RSA)

CONTACTS AND LOCATIONS:
Overall Officials: Are H Stødle, cand. med., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided